CLINICAL TRIAL: NCT02105493
Title: A Novel Approach to Reduce Radial Artery Occlusion After Trans-Radial Catheterization: Post-Procedural/Pre-Hemostasis Intra-Arterial Nitroglycerin
Brief Title: Nitroglycerin Prevents Radial Artery Occlusion
Acronym: NORAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Surya Dharma, MD, PhD, MD, PhD, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NORAO2014
Record Dates: First submitted 2014-02-19; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Injury of Radial Artery
Keywords: Nitroglycerin; Radial Artery Occlusion; Transradial Catheterization
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 500 microgram of Nitroglycerin (Active Comparator): 500 mcg nitroglycerin was given intra-arterially through the sheath at the end of a transradial procedure
  Interventions: Drug: 500 microgram of Nitroglycerin
- Saline 5 mL (Placebo Comparator): 0,9% Saline 5 mL was given intra-arterially through the sheath at the end of a transradial procedure
  Interventions: Drug: Saline 5 mL

INTERVENTIONS:
Drug: 500 microgram of Nitroglycerin — 500 microgram of Nitroglycerin (in 5 mL saline) given intra-arterially through the sheath at the end of transradial procedure
  Other Names: NTG
  Arms: 500 microgram of Nitroglycerin
Drug: Saline 5 mL — Saline 5 mL given intra-arterially through the sheath at the end of transradial procedure
  Other Names: NaCl 0,9% 5mL
  Arms: Saline 5 mL

SUMMARY:
Trans-radial approach (TRA) has becoming popular and widely adopted over the last decade. However, radial artery occlusion (RAO) continues to be one of the limitation of trans-radial access and potentially limits the radial artery as an access site in the future. Several strategies have been used to decrease the incidence of RAO including the use of anticoagulation, maintenance of patency during hemostasis, or shortening the duration of compression. Currently, there is no data whether vasoactive pharmacological therapy such as nitroglycerin administered intra-arterially at the end of the procedure may reduce the incidence of RAO. It is hypothesized that the addition of nitroglycerin (nitric oxide donor) at the end of a TRA procedure may reduce the incidence of RAO.

ELIGIBILITY:
Inclusion Criteria:

* Sequential patients undergoing trans-radial catheterization in the institution will be consented to be randomized to receive either 500 microgram nitroglycerin (Group A) or a placebo (Group B) administered intra-arterially through the sheath at the end of the procedure.

Exclusion Criteria:

* Patients with cardiogenic shock or hemodynamically unstable
* Unable to tolerate nitrates

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1706 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence of radial artery occlusion as confirmed by absence of antegrade flow in vascular high resolution ultrasound | One Day After the Index Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Surya Dharma, MD, PhD, Principal Investigator — National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Derived] Dharma S, Kedev S, Patel T, Sukmawan R, Gilchrist IC, Rao SV. Post-procedural/pre-hemostasis intra-arterial nitroglycerin after transradial catheterization: A gender based analysis. Cardiovasc Revasc Med. 2016 Jan-Feb;17(1):10-4. doi: 10.1016/j.carrev.2015.12.002. Epub 2015 Dec 22. PMID 26797427